CLINICAL TRIAL: NCT03632096
Title: Evaluation of Photobiomodulation in Salivary Production of Patients With Xerostomy Induced by Anti-hypertensive Drugs
Brief Title: Photobiomodulation in Salivary Production of Patients With Xerostomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Malu
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: The sham group will have a simulation of application of the laser, with the device turned off. Because it is an infrared light, it is invisible and this will not induce the patient to notice that the device is turned off. In the group that receives the photobiomodulation the device will have its timer turned off, to avoid the perception of sound difference.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): Patients will receive 3 applications of low intensity light directly in the region of the three pairs of salivary glands already described. The ArGaAl diode laser, DMC 808nm 4J/point equipment will be used. The parameters that will be used are: Laser Diode ArGaAl, DMC, 808nm, 4J per point, continuously and in contact with the irradiated surface, resulting in irradiance of 3571 mW/cm2, distributed as follows: 6 points in each parotid, 2 points in each sublingual (external) and two in each submandibular (internal), totaling 16 extra oral and 4 intra oral, totaling 20 points. The exposure time will be 40s per point, corresponding to 800s per session and 3600s at the end of the four treatment sessions. The radiant exposure will be 142J/cm2. The first application will be after the stimulated collection of saliva and the following applications will be given once a week for another 2 weeks.
  Interventions: Radiation: Photobiomodulation
- Sham group (Sham Comparator): The placebo group will have a simulation of application of the laser, following the same technique as the active group, but with the device turned off. Because it is an infrared light, it is invisible and this will not induce the patient to notice that the device is turned off.
  Interventions: Radiation: Sham

INTERVENTIONS:
Radiation: Photobiomodulation — The parameters are: Laser Diode ArGaAl, DMC, 808nm, 4J per point, continuously and in contact with the irradiated surface, resulting in irradiance of 3571 mW/cm2, distributed as follows: 6 points in each parotid, 2 points in each sublingual (external) and two in each submandibular (internal), totaling 16 extra oral and 4 intra oral, totaling 20 points. The exposure time will be 40s per point, corresponding to 800s per session and 3600s at the end of the four treatment sessions. The radiant exposure will be 142J/cm2.
  Arms: Photobiomodulation group
Radiation: Sham — The sham group will have a simulation of laser application, following the same procedures as the active group, but with the device switched off.
  Arms: Sham group

SUMMARY:
Xerostomia is a quantitative and qualitative alteration of saliva, a symptom present in individuals who make continuous use of medications to control chronic diseases, including hypertension. Difficulties in mastication, swallowing, phonation and palate are present, besides oral burning syndrome, periodontal disease, root caries and bad breath that will interfere in the quality of life, making it difficult to socialize in society. Currently, the methods presented for treatment of xerostomia are palliative, so their use does not consist of an effective treatment. The objective of this study is to evaluate the efficacy of photobiomodulation in the production of saliva in patients with xerostomia induced by antihypertensive drugs. The method consists in the application of the low intensity laser in the three pairs of salivary glands - parotid, submandibular and sublingual. The parameters that will be used are: Laser Diode ArGaAl, DMC, 808nm, 4J per point, continuously and in contact with the irradiated surface, resulting in irradiance of 3571 mW/cm2, distributed as follows: 6 points in each parotid, 2 points in each sublingual (external) and two in each submandibular (internal), totaling 16 extra oral and 4 intra oral, totaling 20 points. The exposure time will be 40s per point, corresponding to 800s per session and 3600s at the end of the four treatment sessions. The radiant exposure will be 142J/cm2. The control group will have a simulation of the application of the laser, with the device turned off. Because it is an infrared light, it is invisible and this will not induce the patient to notice that the device is turned off. In the group that receives the photobiomodulation the device will have its timer turned off, to avoid the perception of sound difference. At the end of the sessions, a sample of saliva will be collected, which will be compared to the initial sample.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients using antihypertensive drugs who present xerostomia;
* Hospitalized in the high-stay unit of the Mandaqui Hospital Complex;
* Patients who sign the free and informed consent form.

Exclusion Criteria:

* Patients with cancer in the oral region;
* Patients receiving radiation therapy;
* Patients with Sjögren's Syndrome;
* Diabetics and those with any type of photosensitivity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-12-10 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Sialometry (measurement of the amount of produced saliva before and after treatment) | One month.
  The patient will be instructed to keep the head forward allowing all saliva to passively pass through the collection tube, resting on the lower lip, for five minutes. In the last second, the patient will be instructed to spit out all the accumulated saliva in the collection tube. The amount of saliva and foam will be evaluated and properly recorded. Then, the dimethicone (removal of the air bubbles) will be used to obtain the final result. At the end of the photobiomodulation sessions a sample of saliva will be collected to be compared to the initial sample. The measurement will be made as follows: milliliters of saliva produced per minute. For stimulate sialometry, a sialogogue will be used. The quantity will be classified as follows: Production of normal saliva: 1.5 to 3.0 ml/minute; Light hyposalivation: from 1.05 to 1.45 ml/minute; Moderate hyposalivation: 0.55 to 1.0 ml/minute; Severe hyposalivation: from 0.05 to 0.50 ml/minute; Sialorrhea: above 3.0 ml/min.

CONTACTS AND LOCATIONS:
Locations (1):
- UniNove, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Varellis MLZ, Goncalves MLL, Pavesi VCS, Horliana ACRT, de Fatima Teixeira da Silva D, Motta LJ, Barbosa Filho VF, Bezerra CDS, Silva FGD, Bussadori SK, Deana AM. Evaluation of photobiomodulation in salivary production of patients with xerostomy induced by anti-hypertensive drugs: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Apr;99(16):e19583. doi: 10.1097/MD.0000000000019583. PMID 32311925